CLINICAL TRIAL: NCT00269620
Title: An Open-Label, Randomized, Multicenter Trial to Evaluate Continuation Rates, Side Effects and Acceptability of NuvaRing Versus OrthoEvra
Brief Title: PARIS or PAtch RIng Study: A Trial to Evaluate NuvaRing Versus OrthoEvra
Acronym: PARIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Organon (Industry)
Responsible Party: Mitchell Creinin, MD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pittirb0503164
Record Dates: First submitted 2005-09-12; First posted 2005-12-23 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Contraception
Keywords: contraceptive vaginal ring; contraceptive patch; oral contraceptives; acceptability
MeSH Terms: interventions — Ethinyl Estradiol; NuvaRing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): OrthoEvra
  Interventions: Drug: ethinyl estradiol/norelgestromin transdermal contraceptive
- 1 (Experimental): NuvaRing
  Interventions: Drug: ethinyl estradiol/etonogestrel vaginal ring

INTERVENTIONS:
Drug: ethinyl estradiol/etonogestrel vaginal ring — vaginal ring for cyclic use (3 weeks in, 1 week out)
  Other Names: Nuvaring
  Arms: 1
Drug: ethinyl estradiol/norelgestromin transdermal contraceptive — contraceptive patch worn for 7 days and replaced for use for 3 consecutive weeks followed by a one-week patch free interval
  Other Names: OrthoEvra
  Arms: 2

SUMMARY:
This is an open-label prospective, multicenter, randomized trial to compare continuation rates into the fourth cycle of women using either the NuvaRing or OrthoEvra. Five hundred women will be recruited at 9 centers nationwide to be randomly assigned to use either the NuvaRing or OrthoEvra for four months. Women must either be on the pill or have recently stopped the pill and be relatively satisfied with oral contraceptive use to qualify for enrollment. Two visits and two phone calls will be required.

DETAILED DESCRIPTION:
The present study is designed primarily to compare continuation rates after three months of use of NuvaRing® and OrthoEvra® in women who had been previously using oral contraceptives. The study attempts to evaluate the possible choices for women who are content with their current or recent method of oral combined hormonal contraception but would be considering a change in their method to a non-daily delivery system. Continuation rates should demonstrate the overall acceptance of both methods as women who find that the method is convenient and has few side effects are likely to continue using the method. Sexual functioning is another important aspect to investigate. The Female Sexual Function Index (FSFI) will be administered to participants along with the planned study questionnaires at the enrollment visit and at the final visit. Additionally, this study will compare side effects, the incidence of bacterial vaginosis, and direct measures of acceptability between the two groups. Efficacy over the three-month study period will also be evaluated; however, since both methods are highly effective and the study is relatively short in duration, the study is not designed to be large enough to detect any differences in efficacy.

This open-label, prospective, multicenter, randomized comparative trial will be conducted in approximately 500 women in the United States who are currently or recently have used a combined oral contraceptive and have no past experience using NuvaRing® or OrthoEvra®. Subjects will be enrolled once they have provided informed consent, had a baseline blood pressure and breast and pelvic examinations, and had negative endocervical testing for gonorrhea and chlamydia. Participants will be randomized to use either NuvaRing® or OrthoEvra® for four continuous cycles beginning with the first day of menses following the enrollment visit. Subjects are to contact the research office by phone to confirm that they initiated the method as instructed. The researchers will contact subjects during the second week of the second cycle of study medication. A final visit will occur during the first week of the fourth cycle of study medication (or sooner if the subject requires or requests early discontinuation). An acceptability questionnaire will be administered at the subject's final visit. This questionnaire has been modified from a questionnaire validated in women using NuvaRing®.

ELIGIBILITY:
Inclusion Criteria:

* Currently or recently (within 3 months of enrollment) using oral contraceptives and content with use.
* In good general health with no contraindications to combined hormonal contraceptive use; premenopausal; and willing to be randomly assigned to use the patch or ring for the next 4 cycles.
* Willing to forego the use of vaginal products and anal intercourse for study duration; if heterosexually active, must be with a single partner for at least the past 3 months and not planning a change during study participation.

Exclusion Criteria:

* Known or suspected pregnancy; hypersensitivity to NuvaRing or OrthoEvra; present or use within 2 months of liver-enzyme-inducing medications or St. John's Wort; breastfeeding currently or within 60 days; abortion or delivery of pregnancy at 15 weeks or greater within 49 days; or abortion within 21 days at 14 weeks or less.
* Previous use of patch or ring for contraception; use of an injectable contraceptive within 6 months; use of an investigational drug within 2 months; or planning a pregnancy within 6 months.
* Diagnosis of gonorrhea or chlamydia at screening, or any vaginal or cervical abnormality that would require colposcopy during the course of the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2005-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
continuation into the fourth cycle | four months

SECONDARY OUTCOMES:
planned continuation after four cycles | four months
compare side effect rates | four months
compare acceptability | four months
evaluate changes in sexual functioning as compared to baseline | four months
compare changes in Nugent's scores (evaluations for bacterial vaginosis [BV]) | four months
evaluate contraceptive efficacy | four months
evaluate number of phone calls and interim visits due to method related problems | four months

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell D Creinin, MD, Principal Investigator — University of Pittsburgh/Magee-Womens Hospital
Locations (10):
- United States (10):
  - UCLA-Harbor, Los Angeles, California
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - Boston University, Boston, Massachusetts
  - Columbia University, New York, New York
  - Oregon Health Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Eastern Virginia Medical School, Norfolk, Virginia
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Result] Creinin MD, Meyn LA, Borgatta L, Barnhart K, Jensen J, Burke AE, Westhoff C, Gilliam M, Dutton C, Ballagh SA. Multicenter comparison of the contraceptive ring and patch: a randomized controlled trial. Obstet Gynecol. 2008 Feb;111(2 Pt 1):267-77. doi: 10.1097/01.AOG.0000298338.58511.d1. PMID 18238962
- [Derived] Gracia CR, Sammel MD, Charlesworth S, Lin H, Barnhart KT, Creinin MD. Sexual function in first-time contraceptive ring and contraceptive patch users. Fertil Steril. 2010 Jan;93(1):21-8. doi: 10.1016/j.fertnstert.2008.09.066. Epub 2008 Oct 31. PMID 18976753